CLINICAL TRIAL: NCT04123743
Title: Efficacy of Extract of Trigonella Foenum-graceum (Fenugreek) as Topical Phytoestrogen in Skin Aging Treatment of Post Menopausal Women : A Study of COL1A1, COL3A1, Skin Thickness, and Skin Wrinkles
Brief Title: Efficacy of Extract of Trigonella Foenum-graceum as Topical Phytoestrogen in Skin Aging Treatment of Post Menopausal Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Shannaz Nadia Yusharyahya, Head of Geriatric Dermatology Division, Department of Dermatovenereology, Faculty of Medicine, Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Skin Aging

STUDY DESIGN:
Intervention Model Description: The participants will be divided into 2 groups, experimental group and control group. Experimental group will get intervention with topical cream containing Trigonella foenum-graceum extract, while control group will get intervention with placebo topical cream. Both experimental and control group will receive Wardah brand facial wash and Parasol sunscreen SPF 33 as part of the assigned intervention as well.The participants will undergo the assigned intervention for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is done to the participants, care providers, investigator, and outcomes assessor in every stage of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will be given topical cream containing Trigonella foenum-graceum extract, Wardah brand facial wash, and Parasol sunscreen SPF 33.
  Interventions: Drug: Trigonella foenum-graceum extract topical cream; Other: Facial Wash; Other: Sunscreen Cream
- Control Group (Placebo Comparator): The control / placebo group will be given placebo topical cream, Wardah brand facial wash, and Parasol sunscreen SPF 33
  Interventions: Other: Facial Wash; Other: Sunscreen Cream; Other: Placebo

INTERVENTIONS:
Drug: Trigonella foenum-graceum extract topical cream — Topical cream containing Trigonella foenum-graceum extract
  Arms: Experimental Group
Other: Facial Wash — Wardah brand facial wash
Other: Sunscreen Cream — Parasol sunscreen cream SPF 33
Other: Placebo — Placebo topical cream
  Arms: Control Group

SUMMARY:
Skin is subjected to intrinsic aging and extrinsic aging. Intrinsic aging is influenced by genetic and hormonal factors. Estrogen has significant role in modulating skin physiology. In post menopausal women, skin aging is accelerated because of hypoestrogenism. Administration of estrogen can delay the process of skin aging. Phytoestrogens are estrogen-like compounds which can be found naturally in plants. The investigators intend to study the efficacy of Trigonella foenum-graceum extract as topical phytoestrogen in skin aging treatment of post menopausal women.

DETAILED DESCRIPTION:
In this double-blinded unmatched randomized controlled trial, the investigators intend to study the efficacy of Trigonella foenum-graceum extract as topical phytoestrogen in skin aging treatment of post menopausal women. The investigators have gathered 21 participants that will be divided into 2 groups, experimental group and control group. Experimental group will get treatment with topical cream containing Trigonella foenum-graceum extract, while control group will get treatment with placebo cream.

The study will be held in esthetic cluster, Kencana Cipto Mangunkusumo Hospital, and radiology cluster, Kencana Cipto Mangunkusumo Hospital from August 2019 until November 2019.

ELIGIBILITY:
Inclusion Criteria:

* Women with minimum 2 years post menopausal and maximum 8 years post menopausal
* Have skin aging problems that manifested as wrinkles on forehead, crow's feet, and nasolabial fold region
* Estradiol level < 30 pg/mL
* Willing to terminate the routine use of facial cream or treatment during the study duration and at least for 30 days before the study commence
* Willing to follow the study protocol and sign the informed consent

Exclusion Criteria:

* Dermatitis in the region of face
* Using oral/topical hormonal supplement in the last 12 months
* Using products containing retinoic acid or it's derivatives in the last 30 days
* Underwent radiotherapy, facelift, dermabrasion, botox, or facial filler procedures in the last 5 years
* Breast lump or other breast abnormality
* History of cancer or malignancy
* Vein thrombosis
* History of hormonal contraception allergy
* History of ovariectomy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Forehead Wrinkles | Change from initial visit VAS at 12 weeks
  Visual Analogue Scale (VAS) to measure wrinkles in the forehead region (Scale 0-8, with 0-2 categorized as mild wrinkling, 3-5 categorized as moderate wrinkling, and 6-8 categorized as severe wrinkling)
Visual Analogue Scale for Crow's Feet Wrinkles | Change from initial visit VAS at 12 weeks
  Visual Analogue Scale (VAS) to measure wrinkles in crow's feet region (Scale 0-6), with 0-2 categorized as mild wrinkling, 3-4 categorized as moderate wrinkling, and 5-6 categorized as severe wrinkling
Visual Analogue Scale for Nasolabial Wrinkles | Change from initial visit VAS at 12 weeks
  Visual Analogue Scale (VAS) to measure wrinkles in nasolabial region (Scale 0-6), with 0-2 categorized as mild wrinkling, 3-4 categorized as moderate wrinkling, and 5-6 categorized as severe wrinkling
High Resolution Ultrasound | Change from initial visit dermis thickness at 12 weeks
  High resolution ultrasound examination in bilateral cheek region to determine dermis thickness (in milimeter).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia